CLINICAL TRIAL: NCT03485729
Title: A Phase II Study of ONC201 in Recurrent or Metastatic Type II Endometrial Cancer
Brief Title: ONC201 in Recurrent or Metastatic Type II Endometrial Cancer Endometrial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated due to a change in the Sponsor's corporate priorities. The decision to terminate the study was not based on any safety concerns.
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Oncoceutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONC012
Record Dates: First submitted 2018-03-25; First posted 2018-04-02 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Endometrial Cancer Recurrent
MeSH Terms: interventions — TIC10 compound

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Patients received 625 mg dordaviprone (ONC201) once weekly on Days 1, 8, and 15 of each 3-week cycle. Patients were required to undergo a biopsy of their tumor one day after their second dose of dordaviprone (ONC201) on Cycle 1, Day 9.
  Interventions: Drug: Dordaviprone (ONC201)
- Arm B (Experimental): Patients received 625 mg dordaviprone (ONC201) once weekly on Days 1, 8, and 15 of each 3-week cycle. Patients were not required to undergo a biopsy of their tumor.
  Interventions: Drug: Dordaviprone (ONC201)
- Arm C (Experimental): Patients received 625 mg dordaviprone (ONC201) twice weekly on consecutive days on Days 1, 2, 8, 9, 15, and 16 of each 3-week cycle. Patients were required to undergo a biopsy of their tumor one day after their fourth dose of dordaviprone (ONC201) on Cycle 1, Day 10.
  Interventions: Drug: Dordaviprone (ONC201)

INTERVENTIONS:
Drug: Dordaviprone (ONC201) — 625 mg dordaviprone (ONC201)

SUMMARY:
This was a Phase 2, Simon two-stage, non-randomized, open-label, 2-arm trial of dordaviprone (ONC201) in women with metastatic or recurrent Type II endometrial cancer who failed at least 1 prior chemotherapy regimen. Patients with histologically confirmed Type II endometrial cancer, including but not limited to serous, clear cell, carcinosarcoma, adenosquamous, and mixed histologies were eligible.

The primary objective of this study was to determine the efficacy of dordaviprone (ONC201) in metastatic type II endometrial cancer.

Note: This study was completed by predecessor company, Oncoceutics, Inc.

DETAILED DESCRIPTION:
This study included 3 arms: Arm A, Arm B, and Arm C. Dordaviprone (ONC201) was to be administered as a dose of 625 mg by mouth, once or twice each week until disease progression, unacceptable toxicity, or if the patient discontinued for any other reason.

For Arm A and Arm B, ONC201 administration occurred on Days 1, 8, and 15 of each 3-week cycle. For Arm C, ONC201 administration occurred on Days 1, 2, 8, 9, and 15, and 16 of each 3-week cycle.

All patients in Arm A had a biopsy of their tumor one day after the second dose of dordaviprone (ONC201) on Cycle 1, Day 9. All patients in Arm C had a biopsy of their tumor one day after the fourth dose of dordaviprone (ONC201) on Cycle 1, Day 10.

Assessments of objective tumor response were conducted using RECIST version 1.1. Safety was assessed through the reporting of adverse events, measurement of vital signs, electrocardiograms, and clinical laboratory results.

Before the study was terminated, a total of 27 patients were enrolled and received at least 1 dose of dordaviprone (ONC201): 10 patients in Arm A, 14 patients in Arm B, and 3 patients in Arm C.

ELIGIBILITY:
Inclusion Criteria:

A patient had to meet all of the following criteria to be eligible to participate in the study:

1. Had histologically confirmed metastatic or recurrent Type II endometrial cancer (serous, clear cell, carcinosarcoma, adenosquamous, and mixed histologies). For patients with tumors that had mixed histologies, the tumor should have had evidence of some tumor cells with Type II endometrial cancer features.
2. Must have had measurable disease, defined as at least 1 lesion that could be accurately measured in at least 1 dimension in accordance with Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
3. Had availability of at least 12 unstained slides from archival formalin-fixed paraffin-embedded (FFPE) tumor tissue. Available archived tissue biopsies were provided for correlative studies.
4. For Arm A and Arm C, patients must have had disease that was amendable to biopsy and must have been willing to provide consent for a tumor biopsy at baseline (within 30 days of beginning ONC201) an at least 1 on-treatment tumor biopsy.
5. Must have had radiographic disease progression after at least 1 line of systemic cytotoxic therapy for metastatic disease or with progression within 12 months of completing adjuvant chemotherapy.
6. Were aged ≥18 years.
7. Had an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
8. Must have had adequate bone marrow, hepatic and renal function, as defined below:

   * Leukocytes: ≥3000/mcL
   * Absolute neutrophil count: ≥1500/mcL
   * Platelets: ≥100,000/mcL
   * Total bilirubin: ≤1.5 upper limit of normal (ULN)
   * Aspartate aminotransferase/Alanine aminotransferase (SGOT/SGPT): ≤2 ULN
   * Creatinine: ≤1.5 ULN OR
   * Creatinine clearance: ≥60 mL/min/1.732 for patients with creatinine levels above ULN calculated using Calvert formula
9. Had a life expectancy of at least 3 months.
10. Had the ability to understand and willingness to sign a written informed consent and Health Insurance Portability and Accountability Act (HIPAA) consent document.
11. Must have been surgically sterile or postmenopausal or must have agreed to use effective contraception during the period of the trial and for at least 90 days after completion of treatment.

Exclusion Criteria:

A potential patient who met any of the following criteria was ineligible to participate in the study:

1. Had any prior treatment with ONC201.
2. Had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who had not recovered from adverse events (AEs) due to agents administered more than 4 weeks earlier.
3. Patients who had not recovered to baseline or Common Terminology Criteria for Adverse Events (CTCAE) Grade ≤2 from related toxicity to all prior therapies were excluded. Patients with non-serious AEs such as alopecia, fatigue, weakness, loss of appetite, and nausea that were non-significant were not excluded.
4. Had any other prior malignancy from which the patient had been disease-free for less than 3 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of any site.
5. Were unable to swallow capsules.
6. Had impairment of gastrointestinal (GI) function or GI disease that may have significantly altered the absorption of ONC201 (uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
7. Were receiving any other investigational agents.
8. Patients with symptomatic brain metastases were excluded. Patients with asymptomatic and treated central nervous system (CNS) metastases may have participated in this trial. The patient must have completed any prior treatment for CNS metastases >28 days prior to study entry including radiotherapy or surgery. Steroids for the treatment of brain metastasis were not permitted, and patients must have been stable off steroid treatment for 4 weeks prior to enrollment.
9. Had uncontrolled intercurrent illness including but not limited to ongoing or active infection. Or any of the following in the 6 months previous to enrollment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, cerebrovascular accident, transient ischemic attack, or symptomatic pulmonary embolism.
10. Had active inflammatory GI disease, chronic diarrhea (unless related to underlying malignancy or prior related treatment) or history of abdominal fistula, GI perforation, peptic ulcer disease, or intra-abdominal abscess within 6 months prior to study enrollment. Gastroesophageal reflux disease under treatment with proton pump inhibitors was allowed.
11. Known human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy.
12. Had active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may have increased the risk associated with study participation or study drug administration or may have interfered with the interpretation of study results, or in the judgement of the Investigator, would have made the patient inappropriate for entry into the study.
13. Were pregnant or breast feeding.
14. Had known history of cardiac arrhythmias including atrial fibrillation, tachyarrhythmias, or bradycardia, unless arrhythmia was controlled and after cardiology had cleared patient to receive ONC201. Was receiving therapeutic agents known to prolong QT interval; however, the use of Zofran was permitted. Had a history of congestive heart failure or myocardial infarction or stroke in the 3 months prior to enrollment.
15. Concomitant use of potent cytochrome P450 (CYP) A4/5 inhibitors or inducers during the treatment phase of the study and within 2 hours prior to starting study drug administration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 27 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Rutgers, The State University of New Jersey, New Brunswick, New Jersey
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm B: Patients received 625 mg of dordaviprone (ONC201) once weekly on Days 1, 8, and 15 of each 3-week cycle. Patients were not required to undergo a biopsy of their tumor.
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C
Started | 10 | 14 | 3
Completed | 0 | 0 | 1
Not Completed | 10 | 14 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Disease progression | 8 | 13 | 1
Not completed — Hospice care | 1 | 0 | 0
Not completed — Poor performance status | 1 | 0 | 0
Not completed — Illness | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Total
Number analyzed (Participants) | 10 | 14 | 3 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 0 | 11
  >=65 years | 4 | 9 | 3 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 3 | 27
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 8 | 13 | 3 | 24
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 1 | 9
  White | 5 | 8 | 2 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Histologically confirmed metastatic or recurrent Type II endometrial cancer [Count of Participants; unit: Participants] | 10 | 14 | 3 | 27

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival Rate at 2 Months
Description: Progression-free survival rate at 2 months was defined as the percentage of participants who exhibited progression-free survival for >8 weeks (>56 days) following treatment initiation; only Arm B participants were analyzed for this outcome.
Time Frame: 2 months (8 weeks); from treatment initiation to 2 months (8 weeks) following treatment initiation
Population: Note that only Arm B participants were planned to be assessed for progression-free survival at 2 months following treatment initiation. Participants in Arm A and Arm C were required to undergo a biopsy of their tumor during the study; participants in Arm B were not. Therefore, including participants in Arm A and Arm C may have represented a biased subset of the overall target population since some sites of metastases may not have been amenable to biopsy.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm B
Number analyzed (Participants) | 14
Participants | 3

ADVERSE EVENTS:
Time Frame: From the time/date of initiation of study treatment through 30 days following cessation of study treatment (32 months)
Description: Note: The progression of cancer under study was not considered an adverse event.
Arm/Group | Arm A | Arm B | Arm C
All-Cause Mortality (participants affected / at risk) | 5/10 | 4/14 | 2/3
Serious Adverse Events (participants affected / at risk) | 7/10 | 4/14 | 3/3
Other Adverse Events (participants affected / at risk) | 10/10 | 14/14 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=10) | Arm B (N=14) | Arm C (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Lung abscess (Infections and infestations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Embolism (Vascular disorders) | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=10) | Arm B (N=14) | Arm C (N=3)
Anaemia (Blood and lymphatic system disorders) | 4 | 6 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 8 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3 | 0
Chills (General disorders) | 0 | 1 | 0
Disease progression (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 6 | 9 | 1
Mucosal inflammation (General disorders) | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 4 | 1
Pain (General disorders) | 2 | 1 | 0
Pyrexia (General disorders) | 1 | 2 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Lung abscess (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 2 | 3 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 2 | 1
Platelet count decreased (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 2 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 4 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 3 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 3 | 2 | 0
Tremor (Nervous system disorders) | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Umbilical haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Embolism (Vascular disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 3 | 0
Lymphoedema (Vascular disorders) | 2 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Note: This study was terminated due to a change in corporate priorities. The decision to terminate the study was not based on any safety concerns with dordaviprone (ONC201).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 12 months of the completion of the Study at all sites, if no publication of the overall multi-center results has been made, institutions are entitled to publish their locally obtained results, provided the Sponsor is given the opportunity to review and comment. Institution publications may be delayed up to an additional 60 days to allow the Sponsor to seek patent protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT03485729/Prot_SAP_000.pdf